CLINICAL TRIAL: NCT05683067
Title: Microcirculation and Vascular Function After Fontan Surgery
Acronym: MICROFON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0860
Record Dates: First submitted 2022-12-12; First posted 2023-01-12 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Congenital Heart Disease
Keywords: Microcirculation; Fontan Procedure; Vascular Function
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fontan Survivors: The investigator will include Fontan survivors between 16-50 years of age for the study.
  Interventions: Other: Hand Held Capillary Microscopy; Other: Mobile 'O' Graph; Other: quality of life using questionnaires
- People operated for congenital heart diseases: The investigator will include people operated for other types of congenital heart diseases such as tetralogy of Fallot, transposition of great arteries between 16 and 50 years of age
  Interventions: Other: Hand Held Capillary Microscopy; Other: Mobile 'O' Graph; Other: quality of life using questionnaires
- Healthy volunteers: The investigator will include healthy volunteers between 16 to 50 years of age for comparison purpose.
  Interventions: Other: Hand Held Capillary Microscopy; Other: Mobile 'O' Graph; Other: quality of life using questionnaires

INTERVENTIONS:
Other: Hand Held Capillary Microscopy — The investigator will visualize the blood vessel appearance, number, and size they have in their hands, feet, and under the tongue. This procedure is non-invasive and will not cause any pain.
Other: Mobile 'O' Graph — The aortic stiffness will be measured non-invasively using a special blood pressure monitor called Mobile 'O' Graph, which is about size of a pocket diary. 24 hour blood pressure monitoring is optional.
Other: quality of life using questionnaires — The investigator will evaluate the quality of life using questionnaires such as EQ-5D-5L questionnaire and the Minnesota Living with Heart Failure Questionnaire (MLHFQ)

SUMMARY:
Fontan Surgery is done for children with only one working lower chamber of the heart called the 'Single Ventricle'. This surgery involves making connections between the two big veins that drain oxygen deficient blood to the heart and the lung artery directly. Fontan patients may develop long-term complications such as reduced heart function or oxygen levels, increased pressure in the veins, liver or kidney problems etc. The reasons for these complications are poorly understood. The small blood vessels in the body or 'microcirculation' are tiny (can be seen only by microscope) and they supply food and oxygen to the tissues. Very little is known about what happens to the microcirculation in adult Fontan survivors . In this study the investigator want to understand why these adult Fontan survivors develop complications by looking at their microcirculation and comparing them with healthy people and those who were operated for other congenital heart diseases. The study will be conducted in East Midlands Congenital Heart Centre, Glenfield Hospital.

Leicester.

DETAILED DESCRIPTION:
In normal heart, there are two working lower chambers where one chamber pumps the blood to the lungs and other chamber pumps the blood to the body. However, some congenital heart conditions have only one working lower chamber of the heart called the 'Single Ventricle'. This condition is often associated with hole between the heart chambers with increased or decreased blood flow to the lungs. This can lead to mixing of blood in the heart with low oxygen levels in the body. The surgery for single ventricle is usually performed in stages starting from the infancy. Fontan surgery is the last stage where the two big veins that return the blood to the heart is connected to the lung artery directly. This surgery improves the oxygen levels in the blood and lessens the burden on the single ventricle. The blood is not pumped to the lungs by the heart but rather enters passively to the lungs through this new surgical connection. Some people operated for Fontan surgery have many short-term and long-term complications such as increased pressure in veins , poor heart function and low oxygen levels in the blood. In particular, the organs below the chest such as kidney, liver and gut are affected, and all of these predict poor outcomes. The reason for these complications are poorly understood.

The small blood vessels in the body or 'microcirculation' are very tiny and are less than 150 microns in diameter. These includes arterioles, capillaries, and venules. Very little is known about the microcirculation in adult Fontan survivors and its association with aortic stiffness, late complications, and quality of life. In this study, The investigators want to look at the blood vessels in adult Fontan survivors, people operated for other congenital heart diseases, and healthy volunteers using a special microscope called Hand Held Capillary Microscopy. The investigators will visualize their blood vessel appearance, number, and size they have in their hands, feet, and under the tongue. This procedure is non-invasive and will not cause any pain. The aortic stiffness will be measured non-invasively using a special blood pressure monitor called Mobile 'O' Graph, which is about size of a pocket diary. 24 hour blood pressure monitoring is optional. The investigator will also collect the information about the quality of life using questionnaires as few studies have shown that the quality of life is affected in adult Fontan survivors and it was associated with poor vascular function. Age matched healthy controls and adults survivors of other congenital heart surgeries will also undergo these tests for comparison purpose. This study will be conducted at East Midlands Congenital Heart Centre, Glenfield Hospital, Leicester.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated for Fontan procedure or other congenital heart conditions
* Patients ≥ 16 - 50 years of age
* Participant/Parents/Guardian or legal representative willing and able to give Informed Consent for participation in the study
* Able (in the Investigators opinion) and willing to comply with all study requirements

Exclusion Criteria:

* Low blood pressure (90/60 mmHg with symptoms or on intravenous inotropes for maintenance of blood pressure)
* Raynaud's disease
* Autoimmune diseases
* Down's syndrome as they have lower risk for vascular anomalies compared with the general population and may have different microvasculature
* Treatment with sympathomimetic drugs
* Atrial fibrillation or any other arrhythmia which might interfere with vascular function assessments.
* Documented peripheral vascular disease
* Skin disorders such as psoriasis or significant eczema
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Tremor or Inability to keep the hand still for 20 minutes.

Note: Patients treated with angiotensin converting enzyme inhibitors or angiotensin receptor inhibitors, beta blockers, vasodilators, diuretics and digoxin will be included in the study as the majority of Fontan survivors are taking one or more of these drugs for optimization of their circulation or for symptom management. Patients treated with anticoagulants and antiplatelets will be included in the study.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In this study, The investigator want to look at the blood vessels and test the vascular function in Fontan survivors, people operated for other congenital heart diseases, and healthy volunteers between 16 and 50 years of age
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
In this study, the investigator want to look at the microcirculation using hand held capillary microscopy in the young and adult Fontan survivors compared to the age matched healthy people and the people operated for other congenital heart surgeries. | One year
  The microcirculation will be studied in the skin of the hands, feet, and the mouth using handheld capillary microscopy

SECONDARY OUTCOMES:
The investigator want to measure the central blood pressure in the young and adult Fontan survivors compared to the age matched healthy people and the people operated for other congenital heart surgeries. | One year
  The central blood pressure, pulse wave velocity, and the augmentation index will be assessed by Mobile O Graph blood pressure monitor
The investigator will measure the functional outcomes in young and adult Fontan survivors using questionnaires and study its relationship with microvascular assessments and vascular function. | One Year
  The functional status will be assessed by Minnesota living with heart failure questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Glenfield Hospital Leicester, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This will be decided soon by the study team